CLINICAL TRIAL: NCT01255124
Title: Study on Dynamic Changes of the Maternal Anti-EV71 and Anti-CVA16 Antibody Levels in Infants and Young Children
Status: Completed | Type: Observational
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Other Study IDs: JSVCT002
Record Dates: First submitted 2010-12-04; First posted 2010-12-07 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Hand, Foot and Mouth Disease; Anti-EV71; Anti-CVA16
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Umbilical cord blood serum and blood serum, Nasopharyngeal swabs, rectal swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Health infants (ClinicalTrials.gov ID: NCT01183611): The subjects participated in the clinical trial 'The Safety and Immunogenicity of Recombinant Hepatitis B Vaccines in the Health Neonates' in 2007 (ClinicalTrials.gov ID: NCT01183611).

SUMMARY:
Hand, Foot and Mouth Disease（HFMD）is an infectious disease in infants and young children caused by enterovirus. There was a great outbreak of HFMD in China, 2008, which brought not only panic to the people, but also huge economic loss. Since 2008, HFMD has become one of the category c infectious diseases in China. Studies showed that Human Enterovirus 71 (EV71) and coxsackievirus A 16 (CVA16) are the most common reasons for this disease. And the investigators are going to develop the vaccines for this disease. There is an urgent need to know the dynamic changes of the maternal anti-EV71 and ant-CVA16 level in infants and young children. In April 2007, the investigators started a clinical trial named 'The Safety and Immunogenicity of Recombinant Hepatitis B Vaccines in the Health Neonates' (ClinicalTrials.gov ID: NCT01183611). In that study the investigators already built a cohort of Health Neonates, followed them and obtained the blood serum on the day 0, 30, 210 and 360 after born. So, based on the cohort and blood serum the investigators got, the investigators plan this study to retrospectively investigate their HFMD histories from birth and follow-up for another year to get the information about the incidence of HFMD. The investigators also plan to assay the maternal anti-EV71 and anti-CVA16 antibodies on the day0 and the dynamic changes of antibodies on 1st month, 7th month (day 210), 1st year (day 360) and on October, 2010.

DETAILED DESCRIPTION:
Hand, Foot and Mouth Disease（HFMD）is a common infectious disease in infants and young children which is caused by enterovirus. HFMD is one of the category c infectious diseases in China. However a group of picornavirus of enterovirus can caused HFMD, including coxsackievirus A (CVA), coxsackievirus B(CVB), Human Enterovirus 71(EV71), Echovirus(ECHO) and so on, EV71 and CVA16 are the most common reason for this disease. This study is carried out to discover dynamic changes of the maternal anti-EV71 and anti-CVA16 antibody in infants and young children from this study.

Infections of Hand, Foot and Month Disease in infants and young children may lead to a certain proportion of serious cases with various complications or death. The primary aim of this study is to find dynamic changes of the maternal anti-EV71 antibody in infants and young children and to provide basic data for the future application of EV71 vaccines. The second aim of this study is to find dynamic changes of the maternal anti- CVA16 antibody levels in infants and young children The third aim of this study is to discover the risk factors of Hand, Foot and Month Disease and to estimate the burden of disease.Hand, Foot and Mouth Disease（HFMD）is a common infectious disease in infants and young children caused by enterovirus. Since 2008, HFMD has become one of the category c infectious diseases in China. However a group of picornavirus of enterovirus can caused HFMD, including coxsackievirus A (CVA), coxsackievirus B(CVB), Human Enterovirus 71(EV71), Echovirus(ECHO) and so on, EV71 and CVA16 are the most common reason for this disease. This study is carried out to discover dynamic changes of the maternal anti-EV71 and ant-CVA16 in infants and young children from this study.

Infections of Hand, Foot and Month Disease in infants and young children may lead to a certain proportion of serious cases with various complications or death. The primary aim of this study is to find dynamic changes of the maternal anti-EV71 in infants and young children and to provide basic data for the future application of EV71 vaccines. The second aim of this study is to find dynamic changes of the maternal anti-CVA16 levels in infants and young children. The third aim of this study is to discover the risk factors of Hand, Foot and Month Disease and to estimate the burden of disease.

ELIGIBILITY:
Inclusion Criteria:

* The subjects participated in the clinical trial named 'The Safety and Immunogenicity of Recombinant Hepatitis B Vaccines in the Health Neonates'in 2007 (ClinicalTrials.gov ID: NCT01183611).
* Written informed consent obtained from the parent(s) of the subject.
* Subjects who the investigator believes will comply with the requirements of the protocol.

Exclusion Criteria:

* Neonatal jaundice requiring systemic treatment.
* Major congenital defects or serious chronic illness.
* Maldevelopment
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population are the health infants born after September 2007 in 6 countries in Jinagsu Province.
Sampling Method: Non-Probability Sample
Enrollment: 1297 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
dynamic changes of the maternal anti-EV71 | from birth to 3 years old
  dynamic changes of the maternal anti-EV71 in infants and young children

SECONDARY OUTCOMES:
dynamic changes of the maternal anti-CVA16 | from birth to 3 years old
  dynamic changes of the maternal anti-CVA16 in infants and young children
incidence of HFMD | from birth to 3 years old
  retrospectively investigate their HFMD histories from birth and follow-up for another year to get the information about the incidence of HFMD.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-cai Zhu, Master, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China